CLINICAL TRIAL: NCT07163247
Title: Effectiveness of Using Pet-Robotic Intervention to Enhance Spontaneous Breathing Trial Success in Intensive Care Unit Patients
Brief Title: Effectiveness of Pet-Robotic Intervention in Intensive Care Unit Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202505120RINC
Record Dates: First submitted 2025-08-24; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Spontaneous Breathing Trial in ICU; Spontaneous Breathing Trial
Keywords: spontaneous breathing trials; Pet-robotic intervention; anxiety; Robot assisted intervention
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic pet (PARO) companionship (Experimental): Participants will receive companionship from a robotic baby seal pet (PARO) during their spontaneous breathing trials. The intervention will be administered continuously throughout the entire duration of the spontaneous breathing trials period or until the participant meets predefined early termination criteria.
  Interventions: Behavioral: Robotic pet (PARO) companionship
- Standard care (No Intervention): Participant in this arm will receive standard care.

INTERVENTIONS:
Behavioral: Robotic pet (PARO) companionship — The intervention is composed of the following components:
  Duration: Robotic pet companionship lasting 30-120 minutes, depending on clinical goals during each spontaneous breathing trial (SBT).
  Preparation and interaction: PARO is introduced 30 minutes before each SBT to establish emotional connection. Study staff will briefly introduce its interactive features, including responding to stroking, gentle tapping, head movements, and eye blinking. Participants may interact freely with PARO during the intervention.
  Assessment: Outcome measurements are conducted during the intervention. If extubated successfully, a semi-structured interview is conducted three days later.
  Early termination: The intervention is stopped if the participant becomes clinically unsuitable for further SBTs or experiences a serious adverse event (e.g., device dislodgement).
  Additional information: After each SBT, PARO is sterilized and stored in a sealed container in the patient's room.
  Other Names: PARO@ICU
  Arms: Robotic pet (PARO) companionship

SUMMARY:
This study aims to develop a novel nursing intervention involving robotic pet companionship to reduce anxiety in patients undergoing spontaneous breathing trials.

DETAILED DESCRIPTION:
This study aims to investigate the effectiveness of pet robotic intervention during spontaneous breathing trials in adult patients admitted to medical intensive care units. The study explores whether this intervention can alleviate patients' anxiety during the weaning process, as well as enhance successful spontaneous breathing trials and facilitate further extubation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older with clear consciousness.
* Mechanical ventilation for more than 72 hours.
* Previously failed the first spontaneous breathing trial and is clinically ready to undergo a second spontaneous breathing trial.

Exclusion Criteria:

* Multidrug-resistant organism infection.
* Requiring airborne infection isolation precautions (e.g., COVID-19).
* Immunodeficiency (absolute neutrophil count < 500 cells/mL).
* Richmond Agitation-Sedation Scale (RASS) less than -1.
* Patient with a tracheostomy.
* Subjects with implanted cardiac devices (e.g., permanent pacemaker, implantable cardioverter defibrillators)
* Known allergy to the fur of the robotic pet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Behavioral responses | Baseline (within 30 minutes prior to each spontaneous breathing trial from Day 1), then every 30 minutes during each spontaneous breathing trial from Day 1 until extubation, intensive care unit discharge, or early termination.
  Behavioral responses will be assessed using the Motor Activity Assessment Score (MAAS). Data will be analyzed as both continuous and categorical variables.
  Continuous variable: mean MAAS score (range 0-6). Categorical variables: Sedated (MAAS 0-2); Cooperative (MAAS = 3); Agitated (MAAS 4-6).
Subjective Psychological response | Baseline (within 30 minutes prior to each spontaneous breathing trial from Day 1), then every 30 minutes during each spontaneous breathing trial from Day 1 of measurement until extubation, intensive care unit discharge, or early termination.
  Measured by using the Visual Analog Scale for Anxiety (VAS-A), ranging from 0 (no anxiety) to 10 (worst possible anxiety).
Objective Psychological Response | During each spontaneous breathing trial from Day 1 of measurement until extubation, intensive care unit discharge, or early termination.
  Crying or anger for more than five minutes (yes/no).

SECONDARY OUTCOMES:
Signs of respiratory distress - heart rate | Every 5 minutes during each spontaneous breathing trial from Day 1 of measurement until extubation, intensive care unit discharge, or early termination.
  Average heart rate measured in beats per minute (bpm).
Signs of respiratory distress - blood pressure | Every 5 minutes during each spontaneous breathing trial from Day 1 of measurement until extubation, intensive care unit discharge, or early termination.
  Average blood pressure measured in millimeters of mercury (mmHg).
Signs of respiratory distress - respiratory rate | Every 5 minutes during each spontaneous breathing trial from Day 1 of measurement until extubation, intensive care unit discharge, or early termination.
  Average respiratory rate measured in breaths per minute.
Signs of respiratory distress - oxygen saturation | Every 5 minutes during each spontaneous breathing trial from Day 1 of measurement until extubation, intensive care unit discharge, or early termination.
  Average peripheral oxygen saturation measured in percent.
Spontaneous breathing trial outcome | After each spontaneous breathing trial from Day 1 of measurement until extubation, intensive care unit discharge, or early termination.
  Completion of spontaneous breathing trial (Yes/No).
Duration of spontaneous breathing trial | After each spontaneous breathing trial from Day 1 of measurement until extubation, intensive care unit discharge, or early termination.
  Total duration of completed spontaneous breathing trial measured in minutes.
Adverse events | From Day 1 of measurement until extubation, intensive care unit discharge, or early termination.
  All adverse events (AEs), serious adverse events (SAEs), and suspected unexpected serious adverse reactions (SUSARs), as defined by Good Clinical Practice (GCP), will be recorded.
Extubation within 24 hours | Within 24 hours from Day 1 of measurement.
  Extubation is defined as removal of the endotracheal tube after the physician's evaluation and confirmation of readiness. Success is defined as removal of the tube within 24 hours and is measured as yes/no.
Experience of using robotic pet | 3 days after extubation.
  A semi-structured interview will be conducted with participants in the experimental arm. The interview will include the following four domains:
  1. Experiences with the spontaneous breathing trials.
  2. Experiences with robotic pet companionship.
  3. Perceived helpfulness of the robotic pet in alleviating anxiety.
  4. Suggestions for future use of the robotic pet.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan